CLINICAL TRIAL: NCT02524912
Title: Methadone Maintenance Outcome Study in Taiwan: 5-year Follow-up
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: NHRITaiwan
Record Dates: First submitted 2015-08-12; First posted 2015-08-17 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-09

CONDITIONS: Heroin Dependence; Sleep Impairment; Mortality; Quality of Life; Treatment Outcome
MeSH Terms: conditions — Heroin Dependence

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
Methadone maintenance treatment (MMT) has been one of the most effective treatment choices for opioid addicts to reduce their heroin use, criminality and spread of HIV. In Taiwan, MMT has been introduced since 2006. To date, more than 30,000 opioid addicts have ever participated in MMT, but only around 10,000 retains in treatment. Outcomes of the ever-treated MMT patients remain unclear. It is crucial to trace the opioid addicts' treatment career, outcomes and unmet treatment needs for the service providers to modify treatment strategy to help these individual to maintain abstinence. Moreover, understanding of the determinants for these subjects' long-term outcomes is important for policy makers to implement realistic policies to motivate the service providers and patients.

From the results of previous research, the research team found that early dropout, defined as stayed in-treatment less than one month, of MMT participants were 14.4%. The rate of maintaining in treatment at 3rd , 6th, and 12th month were 65.7%、51.3% and 33.8%, respectively. Average treatment days for 12-month is 186.9±141.2. This result showed that the effectiveness of the MMT was varied among different facilities. On the other hand, the quality of the MMT can be improved largely through different dimensions. Besides, if one participant can enhance its motivation in staying in-treatment, it could reduce 15% early dropout. Above all, the result also showed that though the quality of life was recorded as improved after MMT, it appeared to be significantly lower than their healthy counterparties. The assessments of health outcomes after participating MMT are rare, but in need. It is necessary to make some modification to improve the effectiveness. Moreover, the evaluation of the needs shall not limit to patients, but also extend to their family members.

Therefore, in this study, the research team plans to probe the dimensions from physical, psychiatric, to social conditions by assessing patients and their family members after treated by MMT for five years. The research team would like to know more about the outcomes of those who attended MMT five years ago, their physical and mental health conditions, also health status of their family members.

ELIGIBILITY:
Inclusion Criteria:

* Attended EC0980203, EC0980209, EC1010102 projects
* Nationality: Taiwan
* 20-year-old and above
* Match the diagnosis of heroin dependence from DSM-IV
* Able to fill out the informed consent

Exclusion Criteria:

* Acute major physical or mental illness (need immediate health care)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included participants in this current study from those who attended our three studies before (IRB approved ID: EC0980203, EC0980209, EC1010102).
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | Five-year

SECONDARY OUTCOMES:
Sleep impairment via Chinese version of the Pittsburgh Sleep Quality Index | One month